CLINICAL TRIAL: NCT00941811
Title: An Explorative, Single Center and Controlled Study to Analyze the Immune Escape Mechanisms of HPV-associated Lesions and to Evaluate the Efficiency and Mechanisms of Imiquimod Treatment of Vulvar Intraepithelial Neoplasias 2/3 (VIN) and Anogenital Warts
Brief Title: Immunevasion of Human Papillomavirus (HPV) in Vulvar Intraepithelial Neoplasia 2/3 and Anogenital Warts and Efficiency and Mechanisms of Imiquimod Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stephan Polterauer, md, Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: _1.0; ISRCTN: 2008-004893-42
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: HPV
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Imiquimod — Local Imiquimod three times weekly for 16 weeks
  Other Names: Aldara

SUMMARY:
The occurance and clinical course of human papillomavirus (HPV)-induced lesions is largely determined by the nature of the cellular immune defense generated. Even tough both genital warts and vulvar intraepithelial neoplasia (VIN) are HPV-associated genital lesions they differ in their risk of malignant progression. Imiquimod (IMQ) is a topically applied Toll-like receptor (TLR) 7 agonist that has been approved for the treatment of superficial (pre-) carcinomas of the skin (basal cell carcinomas, actinic keratosis) and HPV-associated lesions (genital warts). It acts by activation of the immune system exerting anti-tumor and anti-viral properties. The aim of the study is to evaluate the mechanisms of IMQ treatment and to analyze the differences in HPV-affected and non affected tissue at cellular and molecular level as determined by immunofluorescence stainings and real time PCR, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically proven Vulvar Intraepithelial Neoplasia 2/3 and/or anogenital Condyloma acuminata
* Age 18-50
* Informed consent

Exclusion Criteria:

* Malignancy
* Pregnancy
* Therapeutic Immunosupression
* Severe systemic dermatologic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Analysis of Cellular and Molecular Mechanisms of Imiquimod tretament and differences in HPV afeected and non affected tissue at cellular and molecular level | 16 weeks

SECONDARY OUTCOMES:
Proportion of histological and clinical response to therapy after 16 weeks of IMQ therapy | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Georg Stingl, Prof., Principal Investigator — Medical University of Vienna
Locations (1):
- Stephan Polterauer, Vienna, Austria